CLINICAL TRIAL: NCT05072171
Title: Dynamic Responsivity of Inguinal Hernia Scaffold ProFlor Attracts Myogenetic Growth Factors Finalizing the Regeneration of the Herniated Groin
Brief Title: Evidence of Myogenic Growth Factors in 3D Dynamic Inguinal Hernia Scaffold ProFlor
Acronym: HERNIA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Prof. Antonino Agrusa, Associated professor, University of Palermo
Other Study IDs: HERNIA 01_2021
Record Dates: First submitted 2021-09-16; First posted 2021-10-08 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Biopsies from 3D hernia scaffold ProFlor in the short term: 3 patients biopsied 3-5 weeks post implantation of ProFlor
  Interventions: Procedure: Inguinal hernia repair with dynamic prosthesis
- Biopsies from 3D hernia scaffold ProFlor in the midterm: 5 patients biopsied 3-4 months post implantation of ProFlor
  Interventions: Procedure: Inguinal hernia repair with dynamic prosthesis
- Biopsies from 3D hernia scaffold ProFlor in the long term: 4 patients biopsied between 3-4 months post implantation of ProFlor
  Interventions: Procedure: Inguinal hernia repair with dynamic prosthesis
- Biopsies from 3D hernia scaffold ProFlor in the extra long term: 3 patients biopsied more than 3 years after implantation of ProFlor
  Interventions: Procedure: Inguinal hernia repair with dynamic prosthesis

INTERVENTIONS:
Procedure: Inguinal hernia repair with dynamic prosthesis — Tissue specimens excised at the above defined postoperative stages were fixed in neutral-buffered 10% formalin and routinely processed to paraffin wax. Sections (4 μm thick) were cut and stored at room temperature until use. Sections were stained with hematoxylin and eosin (H&E) for histological analysis and Azan trichrome (Bioptica) staining to evaluate muscular tissue in the implant fabric.

SUMMARY:
The study utilizes the same tissue specimens gathered for previous investigations and removed from 15 patients already operated for inguinal hernia, who for different reasons needed additional surgery in the previously operated groin.

DETAILED DESCRIPTION:
Among the individual of investigated the cohort, seven patients underwent groin revision for subsequent hydrocele, 4 for recurrence, and 4 for overlooked ipsilateral multiple hernia protrusions. Made from low weight, large porous polypropylene, ProFlor is composed of a multilamellar cylindrical 3D core, 15 mm thick, with 2 different longitudinal dimensions, 25 or 40 mm. The center of the implant core is connected on one surface to a flat mesh of different width depending on the dimension of the 3D core. This flat part of the device is intended to be deployed to counterface the peritoneal sheath. The 3D core of ProFlor ® is arranged to be compressible on both planes, longitudinal and transversal. Due to its proprietary centrifugal expansion, it can be positioned, fixation free, into the hernia defect for permanent obliteration. ProFlor owns an inherent dynamic responsivity as it contracts and relaxes in accord to the movements of the inguinal floor in which is positioned.

The biopsies were excised from the anterior aspect of the 3D device. It should be noted that once deployed the anterior surface of ProFlor merely faces the external oblique fascia and has no contact with other structures of the groin. Therefore, corruption by host native tissue can be excluded. The biopsies were carried out in ten patients, three in the short term postop. between 3 and 5 weeks, five in the mid-term between 3 and 4 months postop., four in the long-term between 6 and 8 months postop. and the latter three in the extra-long term postop., more than three years after implantation.

ELIGIBILITY:
Inclusion Criteria:

* patients already operated for inguinal hernia with ProFlor, who for different reasons needed additional surgery in the previously operated groin
* ASA score >4

Exclusion Criteria:

* Patients who do not underwent inguinal hernia repair with ProFlor

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Biopsies from ProFlor carried out in 15 patients: 3 in the short term postop. between 3-5 weeks, 5 in the mid-term between 3-4 months postop., 4 in the long-term between 6-8 months postop. and the latter 3 in the extra-long term postop., more than 3 years after implantation
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
assessment of NGF stained areas | 3-5 weeks postop
  evidence in ProFlor of NGF in the short term post implantation
assessment of NGF stained areas | 3-4 months postop.
  evidence of NGF in the midterm post implantation of ProFlor
assessment of NGF stained areas | 6-8 months post implantation
  evidence in ProFlor of NGF in the long term post implantation
assessment of NGF stained areas | >3 years post implantation of ProFlor
  evidence in ProFlor of NGF in the extra long term post implantation
assessment of NGFR p75 stained areas | 3-5 weeks postop
  evidence in ProFlor of NGFR p75 in the short term post implantation
assessment of NGFR p75 stained areas | 3-4 months postop.
  evidence in ProFlor of NGFR p75 in the midterm post implantation
assessment of NGFR p75 stained areas | 6-8 months post implantation
  evidence in ProFlor of NGFR p75 in the long term post implantation
assessment of NGFR p75 stained areas | >3 years post implantation of ProFlor
  evidence in ProFlor of NGFR p75 in the extra long term post implantation

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Agrusa, Professor, Principal Investigator — University of Palermo - Italy

IPD SHARING:
Plan to Share IPD: Undecided